CLINICAL TRIAL: NCT07034768
Title: A Phase 1, 2-Part, Open-Label Study to Evaluate the Pharmacokinetics of a Single Oral Dose of EDG-7500 in Participants With Impaired and Normal Renal Function
Brief Title: A Study to Evaluate EDG-7500 in People With Renal Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EDG-7500-105
Record Dates: First submitted 2025-06-09; First posted 2025-06-24 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Renal Impairments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Volunteers (Experimental)
  Interventions: Drug: EDG-7500
- Severe Renal Impairment (Experimental)
  Interventions: Drug: EDG-7500
- Moderate Renal Impairment (Experimental)
  Interventions: Drug: EDG-7500
- Mild Renal Impairment (Experimental): This arm will only be conducted if deemed necessary based on data in participants with moderate and severe renal impairment
  Interventions: Drug: EDG-7500

INTERVENTIONS:
Drug: EDG-7500 — Single dose of EDG-7500

SUMMARY:
The purpose of this Phase 1 study is to understand and compare the amount of EDG-7500 in the blood after a single dose in participants with different levels of kidney function impairment versus participants with normal kidney function. The safety of EDG-7500 in participants with different levels of kidney function impairment will also be evaluated in this study.

ELIGIBILITY:
Key Inclusion Criteria:

All Participants

* Adult, male or female, 18-75 years of age, inclusive
* Female and male participants must follow protocol-specified contraception guidance
* Continuous non-smoker or light smoker (≤ 5 cigarettes per day or equivalent) for at least 3 months prior to dosing
* BMI ≥ 18.0 and ≤ 40.0 kg/m2 at the screening visit.

Participants with Severe, Moderate and Mild Renal Impairment (RI)

* With the exception of RI and other stable diseases, participant is sufficiently healthy for study participation including the following:

  * Heart rate ≥ 40 bpm and ≤ 110 bpm.
  * QTcF interval ≤ 500 msec and has ECG findings considered normal or not clinically significant.
  * Liver function test including ALT ≤ ULN, AST ≤ ULN, and total bilirubin ≤ 1.5 ULN
* Has impaired renal function as determined by eGFR:

  * eGFR <30 mL/min, not requiring hemodialysis, for participants with severe RI.
  * eGFR ≥30 but <60 mL/min for participants with moderate RI.
  * eGFR ≥60 but <90 mL/min for participants with mild RI.
* Has stable renal function with no clinically significant change in renal status at least 28 days prior to dosing and is not currently or has not been previously on dialysis for at least 1 year.

Participants with Normal Renal Function

* Medically healthy, including the following:

  * Blood pressure ≥ 90/40 mmHg and ≤ 150/95 mmHg
  * Heart rate ≥ 40 bpm and ≤ 100 bpm
  * QTcF interval ≤ 470 msec and has ECG findings considered normal or not clinically significant
  * Liver function test including ALT ≤ ULN, AST ≤ ULN, and total bilirubin ≤1.5x ULN
  * Normal renal function with eGFR ≥ 90 mL/min

Exclusion Criteria:

All Participants

* History or presence of alcohol or drug abuse within the past 2 years prior to dosing.
* Female participant with a positive pregnancy test at the screening visit or at check-in or who is lactating.
* Positive urine or breath alcohol results. Unable to refrain from or anticipates the use of any drugs.
* Positive results for HIV, HBsAg, or HCV.
* Donation of blood or significant blood loss within 56 days prior to the first dosing.
* Plasma donation within 7 days prior to the first dosing.
* Participation in another clinical study within 30 days or within 5 half-lives (if known), prior to dosing.

Participants with Severe, Moderate, and Mild RI (Cohorts 1, 2, and 4)

* History or presence of renal artery stenosis.
* Renal transplant or nephrectomy in ≤ 5 years.
* Diabetes confirmed with HbA1c > 8.5%.

Participants with Normal Renal Function (Cohort 3)

-History of any illness that might confound the results of the study or poses an additional risk to the participant by their participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from time zero to last quantifiable concentration (AUC0-last) | Pre-dose to day 11
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUC0-last)
Area under the curve from time zero to extrapolated infinite time (AUC0-inf) | Pre-dose to day 11
  Area under the plasma concentration time-curve from zero to extrapolated infinite time (AUC0-inf)
Maximum observed plasma concentration (Cmax) | Pre-dose to day 11
Observed plasma concentration at the end of the dosing interval (C24) | Pre-dose to day 11
Time to reach maximum observed plasma concentration (Tmax) | Pre-dose to day 11
Plasma elimination half-life (T1/2) | Pre-dose to day 11
  The time measured for the plasma concentration to decrease by one half.

SECONDARY OUTCOMES:
Amount of unchanged drug excreted in urine from zero to 24 hours post dose (Ae0-24) | From day -1 to day 11
Fraction of drug excreted unchanged in urine (fe) | From day -1 to day 11
Renal clearance | From day -1 to day 11

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No